CLINICAL TRIAL: NCT02878590
Title: Clinical Study for the BONGO Device in the Treatment of Obstructive Sleep Apnea
Brief Title: Clinical Study for the BONGO Device in the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoMed Healthscience Inc. (Industry)
Collaborators: RVW Clinical Consulting (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN-C003
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BONGO DEVICE (Experimental): All participants that qualify will receive the intervention of the Bongo device
  Interventions: Device: BONGO DEVICE

INTERVENTIONS:
Device: BONGO DEVICE — A device to be used for the treatment of mild to moderate obstructive sleep apnea

SUMMARY:
Prospective, non-randomized, open label study

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, open label, single-center clinical study for the BONGO NASAL device for the treatment of obstructive sleep apnea. The study consists of two in laboratory polysomnographic studies and a one two week in home period.

ELIGIBILITY:
Inclusion Criteria:

* • Capacity and willingness to sign informed consent

  * ≥ 21 years of age
  * Diagnosis of mild to moderate OSA (AHI ≥ 5 and AHI ≤ 30) within 12 months of the screening visit with the 3% hypopnea criteria
  * Able to tolerate using the device during a day time trial/acclimation
  * Are currently using CPAP or have been prescribed CPAP and are considered CPAP non-adherent (as per either their CPAP data card and/or verbal confirmation of a diagnosis and unwillingness to use CPAP)

Exclusion Criteria:

* • Nasal deformities

  * Severe nasal allergies
  * Rhinitis or moderate nasal congestion, acute upper respiratory (including nasal, sinus or middle ear) inflammation or infection, or perforation of the ear drum
  * Co-morbid sleep disorders
  * Currently on a hypnotic for insomnia (who have had insomnia for more than a month and take a hypnotic on a daily basis and/or transient insomnia being treated)
  * Uncontrolled or serious illness, including but not limited to: severe breathing disorders including hypercapnic respiratory failure, respiratory muscle weakness, bullous lung disease (as seen in some types of emphysema), bypassed upper airway, pneumothorax, pneumomediastinum, etc.; severe heart disease (including heart failure); or pathologically low blood pressure.
  * Full Face Mask user
  * Mouth breather
  * Pregnant (Female subjects of child bearing age will be asked if they are and/or planning on becoming pregnant during the study; acceptable methods of birth control include birth control pills and barrier method)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: jerrold kram, MD, Principal Investigator — California Center for Sleep Disorders
Locations (1):
- California Center for Sleep Disorders, Alameda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 subjects were enrolled (i.e. given a subject number). 6 subjects did not meet the inclusion / exclusion criteria. 5 subjects did not qualify to use the Bongo device at home.
Groups:
- At Home Bongo Users: Subjects that qualified to use the Bongo at home for a two week period followed by a in-laboratory, overnight polysomnogram (PSG).
Period: Overall Study
Arm/Group | At Home Bongo Users
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All subjects that completed the entire study.
Arm/Group | At Home Bongo Users
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Apnea-Hypopnea Index (AHI)
Description: Obstructive Sleep Apnea (OSA) severity is divided into three categories based on the Apnea-Hypopnea Index (AHI) as follows: Mild (AHI of 5 to 15), Moderate (AHI of 15 to 30), and Severe (AHI > 30). AHI is calculated by dividing the number of events (i.e. Apneas and hypopneas) by the number of hours of sleep. The primary outcome for the study was change in AHI, defined as the difference in AHI between the diagnostic PSG study (baseline with no device) and the final PSG study with the Bongo device for the subjects that completed the entire study.
Time Frame: At Diagnostic Baseline PSG and at Final Treatment PSG with the device
Population: All subjects that completed the entire study.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | At Home Bongo Users
Number analyzed (Participants) | 10
events per hour
  Baseline AHI with no device | 15.7 (6.4)
  AHI with Bongo R1 device | 7.1 (4.2)
  Change in AHI | -8.7 (8.3)
Statistical Analysis 1: Comparison: At Home Bongo Users; Test type: Superiority; p = 0.0093, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: On each subject from their screening visit to their final study termination visit.
Arm/Group | BONGO DEVICE
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BONGO DEVICE (N=23)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 — Subject reported they were not feeling well earlier in the day and had chest discomfort, but was now feeling better and came in at night for the PSG with the device.
Nasal abrasion (Skin and subcutaneous tissue disorders) | 1 — Subject reported that they had a nasal abrasion so they opted to not wear the device one of the days at home. Subject wore the device on subsequent days, including at the PSG with the device with no further reported events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT02878590/Prot_SAP_000.pdf